CLINICAL TRIAL: NCT04493905
Title: The Effects of Anesthetic Techniques on Time to Start of Adjuvant Chemotherapy, and Early- and Late-outcomes Following Surgery for Colorectal Cancer A Prospective, Multicenter, International, Observational, Pragmatic Study
Brief Title: Effects of Anesthetic Techniques on Time to Start of Adjuvant Chemotherapy Following Surgery for Colorectal Cancer
Acronym: ENCORE
Status: Completed | Type: Observational
Sponsor: European Society of Anaesthesiology (Other)
Responsible Party: Sponsor
Other Study IDs: ENCORE
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Neoplasms; Anesthesia; Drug Therapy; Surgery
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer in the world with a high postoperative mortality (2 - 6%) as well as a low 5-year survival (40%). Despite advances in surgery and the use of minimally invasive laparoscopic surgery in recent years and adjuvant chemotherapy after surgery, long-term prognosis has only improved marginally. Epidural analgesia is commonly used as a part of the perioperative management of patients undergoing open, colorectal cancer surgery. Not only does it reduce pain and stress, epidurals have been shown to reduce perioperative inflammation and preserve immunological function, all of which may be beneficial in perioperative tumorigenesis. In several retrospective studies, anesthesia and choice of analgesia have shown to improve long-term survival, but no randomized studies have been published in the literature today. Similarly, the benefits of propofol anesthesia in comparison to inhalational anesthesia have recently been high-lighted in relation to cancer surgery, and many patients today request the use of epidurals, total intravenous anesthesia and loco-regional anesthetic technique during surgery, without clear evidence from prospective studies in the literature. Therefore, the question as to the real benefit of anesthesia technique in postoperative outcomes and tumor recurrence remain unanswered, and skepticism abounds amongst both surgeons and anesthesiologists. It is therefore important to study short- and long-term outcomes in patients undergoing CRC surgery, comparing epidural vs. no epidural or inhalational vs. total intravenous anesthesia. However, prospective, randomized studies are costly, require many patients, and the benefits of choice of anesthesia and analgesia on outcome remain uncertain from the current literature. There is a clear diffusion in practice across the world in the choice of anesthesia for patients undergoing CRC surgery, a lack of evidence in the literature and an absence of guidelines on best practice anesthesia care. We believe that by performing a large, prospective, observational, international, pragmatic study, with low costs, it will be possible to answer some of the important questions pertaining to the choice of anesthesia and analgesia. The clinical trials network at the European Society of Anesthesiology will play an important role in the success of this study.

DETAILED DESCRIPTION:
Primary objective To investigate the effect of anaesthetic technique on:

Short term: time to start of adjuvant chemotherapy in patients planned for RIOT Long term: Time to recurrence (TTR) at 3 years. (please see section 4.2 for details) Secondary objectives 0-30-day postoperative morbidity Length of hospital stay and days at home for 30 days (DAH-30) Adverse events related to oncological treatment (chemotherapy, radiotherapy) Study Subjects Patients with stage I-III colorectal cancer (stratified to stage and type of cancer) scheduled for upfront curative surgery.

Study design Prospective, multicentre, international, observational, pragmatic study Planned sample size 10000 patients from > 200 centres (minimum 40 patients/centre) Inclusion criteria Age > 18 years ASA I-III Scheduled for elective (planned) colorectal cancer surgery for stage I-III (open or minimally invasive) Signed written informed consent when requested by the local Ethics committee Exclusion criteria Uncontrolled renal or liver disease, restrictive (limiting mobility) heart failure or ischemic heart disease (ASA IV-V) Speech, language or cognitive difficulties precluding signing informed consent to participate Stage IV colorectal cancer Primary Outcomes Time to return to intended adjuvant (postoperative) chemotherapy (number of days after surgery) Time to recurrence (TTR) of cancer at 3 years (please see section 4.2 for details) Secondary outcome Percentage of complications within 30 days of surgery as graded by the Clavien-Dindo classification Other adverse events not included in the C-D classification within 30 days Length of hospital stay defined as days from index surgery to arrival at original living facility Days at home for 0-30 days (DAH-30) after index surgery Adverse events related to oncological treatment

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* ASA I-III
* Scheduled for colorectal cancer surgery for stage I-III
* Signed written informed consent

Exclusion Criteria:

* Uncontrolled renal or liver disease, restrictive
* (limiting mobility) heart failure or ischemic heart disease
* Emergency surgery for suspected bowel obstruction from colorectal cancer
* Speech, language or cognitive difficulties
* Stage IV colorectal cancer when only palliative surgery is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for colorectal cancer (stage I-III).
Sampling Method: Probability Sample
Enrollment: 5500 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Time in days from onset of surgery for colorectal cancer (Stage I-III) to first initiation of planned adjuvant chemotherapy | 8 weeks
  time between surgery and start of adjuvant chemotherapy
30-day postoperative morbidity assessed by Clavein-Dindo classification | 30 days
  Evaluation of morbidity 30 days after surgery

SECONDARY OUTCOMES:
Postoperative mortality for 0-30 days | 30 days
  Evaluation of mortality 30 days after surgery
Cancer recurrence or cancer-related death at 90 days, 1, 3 years | 90 days - 1 - 3 years
  evaluation of cncer recurrence or dath at 90 days-1 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD/PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Bell M, Buggy DJ, Brattstrom D, Buchli C, Debouche S, Granath F, Riedel B, Gupta A. The effects of anaesthesia and analgesia on short- and long-term outcomes following colorectal cancer surgery: Protocol for an international, pragmatic, cohort study (ENCORE *). Eur J Anaesthesiol Intensive Care. 2024 Apr 26;3(3):e0051. doi: 10.1097/EA9.0000000000000051. eCollection 2024 Jun. PMID 39916820